CLINICAL TRIAL: NCT05726604
Title: 4D CT Scan With Respiratory Gating Versus 3D CT Scan Concerning Cardiac Dosimetry Assesment for Left Sided Breast Cancers Radiotherapy
Brief Title: 4D CT Scan Versus 3D CT Scan Concerning Cardiac Dosimetry Assesment for Left Sided Breast Cancers Radiotherapy
Acronym: RD3D4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022-A02337-36
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Radiation-Induced Vascular Disease; Left Anterior Descending Coronary Artery Stenosis; Radiotherapy Side Effect; Cardiac Ischemia; Left Sided Breast Cancer; LAD (Left Anterior Descending) Coronary Artery Stenosis
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Coronary Artery Disease; Unilateral Breast Neoplasms; Leukocyte adhesion deficiency type 1; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D CT Scan (No Intervention): Assesment of an usual cardiac dosimetry based on 3D CT scan. Only this dosimetry will be used to treat the patients. Because of the crossover model, patients are included in both arms.
- 4D CT scan with respiratory gating (Experimental): Assesment of an experimental cardiac dosimetry based on 4D CT scan. Not used to treat the patients. Because of the crossover model, patients are included in both arms.
  Interventions: Other: Respiratory gating

INTERVENTIONS:
Other: Respiratory gating — 10 minutes breathing motion monitoring during an additional CT scan to establish a more accurate cardiac and LAD dosimetry compared to reality
  Other Names: breathing motion monitoring
  Arms: 4D CT scan with respiratory gating

SUMMARY:
To establish if the cardiac radiation dose assesment is well aproximated with routine 3D CT scan compared to 4D CT experimental scan with respiratory gating (breath motion monitoring). The study population relates to left side breast cancers female patients that require a radiation therapy treatment.

DETAILED DESCRIPTION:
As a standard of care, the postoperative breast cancers radiation therapy is generally based on a 3 dimensions CT scan that does not incorporate the breathing motion by definition.

Meanwhile, the patients must commonly receive the treatment in free motion breathing condition.

More of that, the Cardiac dose, especially the LAD (left anterior descending artery) dose has been established as the main cause of radiation induced ischemic heart disease (RIHD) and should be consider in the first place.

In more concrete terms, the higher the LAD dose is, the greater the RIHD relates: arise the LAD dose by 1 Gy means a 7.4% higher risk to cause a RIHD during the next 5 years.

That being said, to determine if the cardiac dosimetry and the dose-volume histograms (specifically for the left side breast cancer treatments including or not the internal mammary artery) obtained from a 3D CT scan reflect well or not the reality (which is widely subject to the breathing motion).

Finally, because it has been established that a 4D CT scan can monitor the breathing motion, it seems definitely interesting to compare it with the average 3D CT scan to address this concern.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yo
2. Sex=female
3. Patients diagnoses with a left side breast cancer for which a radiation therapy is indicated and confirmed in a multidisciplinary consultation meeting.
4. Be able to understand and give her personal free consent, no judicial protection measure.
5. Written or oral consent, in compliance with the clinical investigation rules and regulation.
6. Patient affiliated with social security system
7. Treatment expected to be realized in Saint Quentin Hospital

Exclusion Criteria:

1. Patient < 18 yo
2. Pregnant women.
3. Breastfeeding women.
4. Consent not given
5. Claustrophobia
6. Incapacited subject or judicial protection measure
7. Other research with exclusion period time ongoing
8. All the inclusion criteria not met

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
3D LAD mean dose vs 4D LAD mean dose | 1 week
  To determine if the mean LAD (left anterior descending artery) dose significantly changes statistically between an usual 3D CT scan versus a 4D CT with breathing motion monitoring (10 breathing phases are monitored).
  Based on stastical test with 95% confidence intervals, to evaluate if there is a significant difference between 4D CT LAD mean dose and 3D CT LAD mean dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Quentin Hospital, Saint-Quentin, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Radiation-Induced CAD: Incidence, Diagnosis, and Management Outcomes, American College of Cardiology 2018, Borges et al — https://www.acc.org/latest-in-cardiology/articles/2018/05/24/01/44/radiation-induced-cad
- See also: Risk of Ischemic Heart Disease in Women after Radiotherapy for Breast Cancer, N England J Med 2013, Darby et al — https://doi.org/10.1056/NEJMoa1209825
- See also: Radiation-induced heart disease: a review of classification, mechanism and prevention, Int J Biol Sci.2019 , Wang et al — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6775290/
- See also: " Comparing whole heart versus coronary artery dosimetry in predicting the risk of cardiac toxicity following breast radiation therapy" Red Journal 102, Sa Patel et al — https://doi.org/10.1016/j.ijrobp.2018.06.091
- See also: Delineation of target volumes and organs at risk in adjuvant radiotherapy of early breast cancer: national guidelines and contouring atlas by the Danish Breast Cancer Cooperative Group" Acta Oncologica 2013, Nielsen et al — https://pubmed.ncbi.nlm.nih.gov/23421926/
- See also: Tangential Field Radiotherapy for Breast Cancer-The Dose to the Heart and Heart Subvolumes: What Structures Must Be Contoured in Future Clinical Trials? Front Oncol 2017, Duma et al. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5474560/